CLINICAL TRIAL: NCT01283763
Title: ITIC2 Trial - Topical Imiquimod Versus Conization to Treat Cervical Intraepithelial Neoplasia: Randomised Controlled, Non-inferiority Trial
Brief Title: Topical Imiquimod Versus Conization to Treat Cervical Intraepithelial Neoplasia
Acronym: ITIC2
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: poor recruitment
Sponsor: Medical University of Vienna (Other)
Collaborators: Medical University of Graz (Other); Medical University Innsbruck (Other); Krankenhaus Barmherzige Schwestern Linz (Other); Salzburger Landeskliniken (Other)
Responsible Party: Principal Investigator, Stephan Polterauer, Ass.Prof. MD, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ITIC2
Record Dates: First submitted 2011-01-21; First posted 2011-01-26 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: Cervical Intraepithelial Neoplasia
Keywords: Cervical Intraepithelial Neoplasia, Imiquimod, conization
MeSH Terms: conditions — Uterine Cervical Dysplasia | interventions — Imiquimod; Conization

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Topical Imiquimod (Experimental): 16 weeks topical Imiquimod
  Interventions: Drug: Topical Imiquimod
- Conization (Active Comparator): Large loop excision of the transformation zone
  Interventions: Procedure: Conization

INTERVENTIONS:
Drug: Topical Imiquimod — 16 weeks
  Other Names: Aldara®
  Arms: Topical Imiquimod
Procedure: Conization — Large loop excision of the transformation zone
  Arms: Conization

SUMMARY:
The purpose of this study is to investigate the non-inferiority of a topical Imiquimod therapy in patients with persistent CIN 2/3 when compared to standard therapy, i.e. conization A randomized, controlled, non-inferiority AGO-Austria trial

DETAILED DESCRIPTION:
Background: Alternatives to surgery are needed for the treatment of cervical intraepithelial neoplasia (CIN). CIN is associated with persistent human papillomavirus (HPV) infection and is known to be a potential precursor of cervical cancer. The incidence of CIN has been increasing during the last decades, especially among young women. Patients diagnosed with (persistent) high-grade CIN (CIN2/3) are treated with conization. Conization can be regarded as a safe procedure but peri- and postoperative complications (infections, bleeding, preterm birth) occur. This raises the need for a conservative treatment alternative for patients with high-grade CIN. Preliminary data: Imiquimod (IMQ), a toll-like receptor 7 agonist, is an immune modulating substance approved for the therapy of superficial skin lesions (e.g. basalioma, actinic keratosis) and HPV associated disease (e.g. anogenital condylomata acuminata and vulvar intraepithelial neoplasia). In a randomized, placebo-controlled phase II trial, we previously showed that topical IMQ therapy is an efficacious and feasible treatment for selected patients with CIN 2/3. Methods: In the present open, randomized, non-inferiority trial 500 women with CIN 2/3 will be included. This non-profit, patient-oriented clinical research project will be conducted as an Austrian Gynecologic Oncology Group (AGO-Austria) trial. Participants will be randomized to either 16 weeks treatment with topical IMQ (new treatment) or to standard therapy i.e. conization (active control). This study investigates the non-inferiority of the new treatment, compared to surgical standard treatment. The primary endpoint is the rate of successful treatment, defined as negative HPV test result six months after treatment start. Six months after start of therapy the primary study endpoint is assessed using HPV genotyping. In addition clinical examinations including colposcopy, HPV genotyping, cytology, and if indicated colposcopy-guided biopsies of the uterine cervix will be performed. In addition, rates of CIN persistence/recurrence 6, 12, 18, and 24 months after start of the treatment and rates of negative HPV test results 12 and 24 months after start of the treatment will be evaluated in both treatment groups.

Rationale: The need for a conservative treatment modality for patients diagnosed with CIN is obvious, as many young women need surgical treatment. In this randomized controlled, trial we will investigate the non-inferiority of a topical IMQ treatment compared to surgical standard treatment in selected patients diagnosed with CIN 2/3.

ELIGIBILITY:
Inclusion criteria:

1. Women aged ≥18 years diagnosed with histologically verified CIN 3 and women aged ≥ 30 years diagnosed with CIN 2
2. Satisfactory colposcopy
3. Signed informed consent
4. Negative pregnancy test
5. Appropriate contraception method for fertile women during active study period
6. Adequate compliance

Exclusion criteria:

1. Adenocarcinoma in situ
2. History of previous conization
3. Malignant disease at the time of inclusion
4. Colposcopy suspicious for invasive disease
5. Pregnancy and lactation period
6. Known allergy or intolerance to IMQ
7. Contraindications to conization or IMQ
8. Symptoms of a clinically relevant disease
9. Known HIV infection
10. Evidence of a clinically significant immunodeficiency
11. Current, reported participation in another experimental, interventional protocol

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2013-05; Primary Completion 2017-09 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
HPV clearance | 6 months after treatment completion
  non-inferiority of experimental treatment (Imiquimod) to active control (conization)

SECONDARY OUTCOMES:
Rates of CIN remission/regression and/or CIN persistence/regression after treatment | 6, 12, and 24 months after treatment completion
  Histologic outcome
HPV clearance | 12 and 24 months after treatment completion

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Polterauer, MD, Principal Investigator — Medical University of Vienna; Stephan Polterauer, MD, Study Director — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria, Austria

REFERENCES:
- [Derived] Polterauer S, Reich O, Widschwendter A, Hadjari L, Bogner G, Reinthaller A, Joura E, Trutnovsky G, Ciresa-Koenig A, Ganhoer-Schimboeck J, Boehm I, Berger R, Langthaler E, Aberle SW, Heinze G, Gleiss A, Grimm C. Topical imiquimod compared with conization to treat cervical high-grade squamous intraepithelial lesions: Multicenter, randomized controlled trial. Gynecol Oncol. 2022 Apr;165(1):23-29. doi: 10.1016/j.ygyno.2022.01.033. Epub 2022 Feb 15. PMID 35177279
- See also: Medical University of Vienna — http://www.meduniwien.ac.at